CLINICAL TRIAL: NCT01511276
Title: The Effects of Equivalent Weight Loss With or Without Exercise Training on Breast Cancer Risk Biomarkers in Postmenopausal Women: the SHAPE-2 Study
Brief Title: The Effects of Equivalent Weight Loss With or Without Exercise Training on Breast Cancer Risk (SHAPE-2)
Acronym: SHAPE-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, E.M. Monninkhof, PhD, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 11-465
Record Dates: First submitted 2012-01-12; First posted 2012-01-18 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer Risk
Keywords: Breast cancer; Sex hormones; Physical activity
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Analyses of the blood assays and MRI data were masked.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Diet-induced weight loss (Experimental): The diet-induced weight loss group will follow a calorie restricted diet. They are asked to keep their habitual sedentary lifestyle. The aim of this group is to loose 5-6 kg of body weight in 14 weeks time.
  Interventions: Behavioral: Diet
- Mainly exercise induced weight loss (Experimental): Participants in the exercise- plus diet-induced weight loss group are enrolled in an exercise programme. Next to the exercise programme, they will follow a calorie restricted diet.
  The aim of this group is to loose 5-6 kg of body weight in 14 weeks time.
  Interventions: Behavioral: Mainly exercise induced weight loss
- Control, stable weight (No Intervention): The control group is asked to follow a baseline isocaloric diet and to not change their habitual sedentary lifestyle.

INTERVENTIONS:
Behavioral: Diet — Energy restricted diet, according the national guidelines for healthy nutrition, creating a mean energy deficit of 500 kCal/day.
  Arms: Diet-induced weight loss
Behavioral: Mainly exercise induced weight loss — Exercise programme of 2 hours per week fitness containing endurance and resistance training. And 2 hours of Nordic Walking. Equivalent to an energy expenditure of 350 kCal/day.
  Next to the exercise programme participants will follow an energy restricted diet according to the national guidelines of healthy nutrition creating an extra energy deficit of 250 kCal/day.
  Arms: Mainly exercise induced weight loss

SUMMARY:
Physical inactivity and overweight are two accepted risk factors for breast cancer. However, because of their correlation it is not clear which is most relevant to risk. The investigators now set out to study whether physical activity in addition to weight loss by diet only, affects sex hormone levels, known to be related to breast cancer risk.

In the SHAPE-2 study 250 healthy overweight/obese and physically inactive women are randomly allocated to a diet-induced weight loss group, a combined exercise- and diet-induced weight loss group or a control group. The aim of the first two intervention groups is to loose 5-6 kg of bodyweight, either by dieting or mainly by increased physical activity. Measurements are performed at baseline and after 21 weeks, the end of the study period.

The aim of this study is to provide insight into the effect of weight loss mainly driven by exercise compared to equivalent weight loss due to nutritional calorie restriction on breast cancer biomarkers.

DETAILED DESCRIPTION:
Postmenopausal women who are sedentary or overweight, have an increased breast cancer risk. It is suggested that these two factors mediate breast cancer risk mainly through sex hormone-related pathways. However, an inactive lifestyle and obesity are highly correlated and it is not clear which is most relevant to risk.

Literature shows that weight loss/ fat loss reduces postmenopausal sex hormone levels, but the question is if there is an additional beneficial effect on hormones of reaching this weight loss by physical activity instead of nutritional interventions.

In this three-armed, two-center intervention study, 250 sedentary postmenopausal women who are aged 50-69 years will first enter a run-in period of 5 weeks. During this period, all participants get a diet, adapted to the guidelines for healthy nutrition, meeting their energy expenditures to maintain stable weight. After this run-in phase they are randomly allocated to a (1) diet induced weight loss group, (2) a combined exercise and diet induced weight loss group or (3) a control group. Participants allocated to the dietgroup will get a calorie restricted diet of -500 kCal/day, they will remain their habitual exercise pattern. Participants in the combined group will follow an exercise programme (combined endurance and strength) of 4 hours of sports per week with an average energy expenditure of 350 kCal/day and a, less strict. And a calorie restricted diet of -250 kCal/day. The aim of both intervention groups is to loose 5-6 kg of body weight during the 14 week intervention period. Participants in the control group are requested to retain the baseline diet and their habitual exercise pattern. Primary study parameters measured at baseline and after 21 weeks are: serum concentrations of endogenous estrogens, endogenous androgens and sex hormone binding globulin. Other study parameters include: body fat distribution, amount of total and abdominal fat, weight, BMI, physical fitness, blood pressure and lifestyle factors.

The aim of this study is to provide insight into the effect of weight loss mainly driven by exercise compared to equivalent weight loss due to nutritional calorie restriction on breast cancer biomarkers. Furthermore, we are specifically interested whether weight loss mainly due to physical exercise induces greater amounts of fat loss (total and abdominal) and subsequently results in more favourable effects on these hormones compared to equivalent diet-induced weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 50-69 years of age
* Postmenopausal (>12 months after last menses)
* BMI 25-35 kg/m2
* Sedentary (<2 hours per week of at least moderately intensive activities (>4 MET))
* Willing to be randomly assigned to one of the three study arms
* Informed consent to participate in all screening and study activities.

Exclusion Criteria:

* Presently using sex-hormones

  * Maintenance use of corticosteroids
  * Suffering cancer (in medical history) except for non-melanoma skin cancers
  * Suffering type II diabetes mellitus or other endocrine related diseases
  * Smoking
  * Alcohol or drug abuse
  * Any disorder that might impede participation in the exercise programme
  * Following, or the intention to follow, a structured weight loss programme elsewhere

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
serum sex hormone levels | 21 weeks
  Estradiol (total, free), estrone, testosterone, sex hormone binding globulin.

SECONDARY OUTCOMES:
anthropometrics and physical fitness. | 21 weeks
  BMI, weight, waist- and hip-circumference, total body fat (DEXA scan), abdominal fat (subcutaneous and visceral, MRI-abdomen) and physical fitness (maximal exercise capacity test by the ramp protocol).

CONTACTS AND LOCATIONS:
Overall Officials: evelyn Monninkhof, PhD, Principal Investigator — UMC Utrecht, Julius Center
Locations (2):
- Netherlands (2):
  - Medisch Spectrum Twente, Enschede, Overijssel
  - UMC Utrecht, Utrecht

REFERENCES:
- [Background] van Gemert WA, Iestra JI, Schuit AJ, May AM, Takken T, Veldhuis WB, van der Palen J, Wittink H, Peeters PH, Monninkhof EM. Design of the SHAPE-2 study: the effect of physical activity, in addition to weight loss, on biomarkers of postmenopausal breast cancer risk. BMC Cancer. 2013 Aug 23;13:395. doi: 10.1186/1471-2407-13-395. PMID 23972905
- [Result] van Gemert WA, van der Palen J, Monninkhof EM, Rozeboom A, Peters R, Wittink H, Schuit AJ, Peeters PH. Quality of Life after Diet or Exercise-Induced Weight Loss in Overweight to Obese Postmenopausal Women: The SHAPE-2 Randomised Controlled Trial. PLoS One. 2015 Jun 1;10(6):e0127520. doi: 10.1371/journal.pone.0127520. eCollection 2015. PMID 26029921
- [Result] van Gemert WA, Schuit AJ, van der Palen J, May AM, Iestra JA, Wittink H, Peeters PH, Monninkhof EM. Effect of weight loss, with or without exercise, on body composition and sex hormones in postmenopausal women: the SHAPE-2 trial. Breast Cancer Res. 2015 Sep 2;17(1):120. doi: 10.1186/s13058-015-0633-9. PMID 26330303
- [Result] van Gemert WA, May AM, Schuit AJ, Oosterhof BY, Peeters PH, Monninkhof EM. Effect of Weight Loss with or without Exercise on Inflammatory Markers and Adipokines in Postmenopausal Women: The SHAPE-2 Trial, A Randomized Controlled Trial. Cancer Epidemiol Biomarkers Prev. 2016 May;25(5):799-806. doi: 10.1158/1055-9965.EPI-15-1065. Epub 2016 Feb 16. PMID 26908432
- [Result] de Roon M, van Gemert WA, Peeters PH, Schuit AJ, Monninkhof EM. Long-term effects of a weight loss intervention with or without exercise component in postmenopausal women: A randomized trial. Prev Med Rep. 2016 Dec 9;5:118-123. doi: 10.1016/j.pmedr.2016.12.006. eCollection 2017 Mar. PMID 27981025
- [Derived] van Gemert WA, Peeters PH, May AM, Doornbos AJH, Elias SG, van der Palen J, Veldhuis W, Stapper M, Schuit JA, Monninkhof EM. Effect of diet with or without exercise on abdominal fat in postmenopausal women - a randomised trial. BMC Public Health. 2019 Feb 11;19(1):174. doi: 10.1186/s12889-019-6510-1. PMID 30744621